CLINICAL TRIAL: NCT02639429
Title: The Efficacy of Transcervical Foley Balloon Plus Vaginal Misoprostol Versus Vaginal Misoprostol Alone For Cervical Ripening In Nulliparous Obese Women: A Randomized, Comparative Effectiveness Trial
Brief Title: Cervical Ripening for Obese Women: A Randomized, Comparative Effectiveness Trial
Acronym: CROWN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Mesk A.Jawad Alrais, Clinical Resident, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-15-0895
Record Dates: First submitted 2015-12-15; First posted 2015-12-24 (Estimated); Results first posted 2019-08-26 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Obesity; Labor Induction; Cesarean Delivery
MeSH Terms: conditions — Obesity | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combined approach: Foley Balloon + Vaginal Misoprostol (Experimental): These women will receive vaginal misoprostol per standard protocol at 25 micrograms every 4 hours. In addition, a 26 Fr-Foley balloon catheter will be inserted by routine clinical standards. The Foley will be inserted through the internal cervical os, filled with 60 mL of normal saline, and then pulled snugly against the internal os. The catheter of the Foley will be taped to the patient's inner thigh under gentle traction. If the Foley is unable to be placed, the patient will be reexamined in 1 hour and placement will be reattempted if Bishop's score is still 6 or less by the healthcare provider. When the Foley balloon had fallen out or had to be removed because 12 hours have passed since insertion as per protocol, further management of labor will be left at the discretion of the labor team.
  Interventions: Device: Foley Balloon + Vaginal Misoprostol
- Single approach: Vaginal Misoprostol only (Active Comparator): These women will receive 25 micrograms of misoprostol per vagina every 4 hours. Once the cervix becomes favorable (Bishop score > 6), misoprostol administration will be discontinued. Further management will be left at the discretion of the labor team.
  Interventions: Drug: Vaginal Misoprostol

INTERVENTIONS:
Drug: Vaginal Misoprostol
  Other Names: Cytotec
  Arms: Single approach: Vaginal Misoprostol only
Device: Foley Balloon + Vaginal Misoprostol
  Arms: Combined approach: Foley Balloon + Vaginal Misoprostol

SUMMARY:
Obese pregnant women (BMI ≥ 30 kg/m2) are more likely than their normal-weight counterparts to require induction of labor because of increased rates of obstetric complications including pregnancy related hypertensive disorders, diabetes, and prolonged gestations. Several studies have shown that obese women experience increased labor duration and oxytocin needs when compared to normal-weight women. This in turn results in increased rates for unplanned cesarean delivery (CD) as a result of failed induction of labor (IOL), arrest disorders and non-reassuring fetal heart rate tracing, that is dose-dependent with increasing class of obesity. The investigators hypothesize that obese pregnant women and unfavorable cervix (Bishop score ≤ 6), IOL ≥ 24 weeks gestation using the Foley balloon plus vaginal misoprostol will result in reduced cesarean delivery rates when compared to vaginal misoprostol alone.

DETAILED DESCRIPTION:
Nulliparous pregnant women at ≥ 32 weeks' gestation admitted to labor and delivery for IOL and who meet the inclusion and exclusion criteria will be approached by the research staff. Group 1 will be composed of women allocated to the Foley balloon plus misoprostol. These women will receive vaginal misoprostol per standard protocol at 25 micrograms every 4 hours. In addition, a 26 Fr-Foley balloon catheter will be inserted by routine clinical standards. The Foley will be inserted through the internal cervical os, filled with 60 mL of normal saline, and then pulled snugly against the internal os. The catheter of the Foley will be taped to the patient's inner thigh under gentle traction. If the Foley is unable to be placed, the patient will be reexamined in 1 hour and placement will be reattempted if Bishop's score is still 6 or less by the healthcare provider. When the Foley balloon had fallen out or had to be removed because 12 hours have passed since insertion as per protocol, further management of labor will be left at the discretion of the labor team.

Group 2 will be composed of women allocated to vaginal misoprostol-only. These women will receive 25 micrograms of misoprostol per vagina every 4 hours. Once the cervix becomes favorable (Bishop score > 6), misoprostol administration will be discontinued. Similarly, further management will be left at the discretion of the labor team.

In both groups, if IV oxytocin is indicated, it will be withheld until 4 hours after the last dose of misoprostol to prevent uterine hyperstimulation. Other aspects of labor management will be similar for both groups, including continuous electronic fetal monitoring with external Doppler device or fetal scalp electrode. Uterine contraction assessment will be performed with either an external tocodynamometer or an intrauterine pressure catheter.

ELIGIBILITY:
Inclusion Criteria

* Nulliparous women aged 18 or above
* BMI ≥ 30 at the time of labor induction
* Singleton gestation
* Cephalic presentation (includes successful external cephalic version)
* Intact fetal membranes
* Unfavorable cervix (Bishop score of ≤ 6)
* Gestational age ≥ 32 weeks

Exclusion Criteria

* Patient not candidate for IOL with misoprostol as deemed by the treating physician
* Multiple gestation
* Major fetal anomalies
* Fetal demise

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2016-01; Primary Completion 2018-06-24 (Actual); Study Completion 2018-06-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas Health Science Center, Houston, Texas, United States

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264
- [Derived] Viteri OA, Tabsh KK, Alrais MA, Salazar XC, Lopez JM, Fok RY, Chauhan SP, Sibai BM. Transcervical Foley Balloon Plus Vaginal Misoprostol versus Vaginal Misoprostol Alone for Cervical Ripening in Nulliparous Obese Women: A Multicenter, Randomized, Comparative-Effectiveness Trial. Am J Perinatol. 2021 Aug;38(S 01):e123-e128. doi: 10.1055/s-0040-1708805. Epub 2020 Apr 16. PMID 32299108

RESULTS

PARTICIPANT FLOW:
Groups:
- Combined Approach: Foley Balloon + Vaginal Misoprostol: These women will receive vaginal misoprostol per standard protocol at 25 micrograms every 4 hours. In addition, a 26 Fr-Foley balloon catheter will be inserted by routine clinical standards. The Foley will be inserted through the internal cervical os, filled with 60 mL of normal saline, and then pulled snugly against the internal os. The catheter of the Foley will be taped to the patient's inner thigh under gentle traction. If the Foley is unable to be placed, the patient will be reexamined in 1 hour and placement will be reattempted if Bishop's score is still 6 or less by the healthcare provider. When the Foley balloon had fallen out or had to be removed because 12 hours have passed since insertion as per protocol, further management of labor will be left at the discretion of the labor team.
  Foley Balloon + Vaginal Misoprostol
- Single Approach: Vaginal Misoprostol Only: These women will receive 25 micrograms of misoprostol per vagina every 4 hours. Once the cervix becomes favorable (Bishop score > 6), misoprostol administration will be discontinued. Further management will be left at the discretion of the labor team.
  Vaginal Misoprostol
Period: Overall Study
Arm/Group | Combined Approach: Foley Balloon + Vaginal Misoprostol | Single Approach: Vaginal Misoprostol Only
Started | 113 | 123
Completed | 113 | 123
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combined Approach: Foley Balloon + Vaginal Misoprostol | Single Approach: Vaginal Misoprostol Only | Total
Number analyzed (Participants) | 113 | 123 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (5.8) | 23.4 (6.1) | 24.3 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 123 | 236
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Amercian | 25 | 26 | 51
  Caucasian | 14 | 15 | 29
  Hispanic | 68 | 74 | 142
  Other | 6 | 8 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 113 | 123 | 236
Gestational Age [Mean (Standard Deviation); unit: weeks] | 38.7 (5.2) | 38.6 (5.4) | 38.6 (5.4)
Number of participants who are married [Count of Participants; unit: Participants] | 64 | 67 | 131
Number of participants who had prenatal care [Count of Participants; unit: Participants] | 110 | 121 | 231
Number of participants with government subsidized insurance [Count of Participants; unit: Participants] | 60 | 73 | 133
Number of participants with hypertensive disease [Count of Participants; unit: Participants] | 60 | 62 | 122
Number of participants with diabetes in pregnancy [Count of Participants; unit: Participants] | 20 | 24 | 44
Body Mass index [Mean (Standard Deviation); unit: kg/m^2] | 38.9 (10.3) | 37.7 (9.6) | 38.3 (10.0)
Bishop score [Median (Inter-Quartile Range); unit: units on a scale] — Bishop score, also known as cervix score, is a pre-labor scoring system to assist in predicting whether induction of labor will be required. Score ranges from 0 to 13. A score of 5 or less suggests that labor is unlikely to start without induction. A score of 9 or more indicates that labor will most likely commence spontaneously. Scores between 5 and 9 require additional consideration and professional judgement for clinical management.
  units on a scale | 3 [2 to 4] | 3 [2 to 5] | 3 [2 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Need for Cesarean Delivery
Time Frame: Induction to delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Approach: Foley Balloon + Vaginal Misoprostol | Single Approach: Vaginal Misoprostol Only
Number analyzed (Participants) | 113 | 123
Participants | 51 | 53

2. Secondary Outcome: Indication for Cesarean Delivery
Description: Categories of Indications for Cesarean Delivery:
  1. = Cephalopelvic disproportion
  2. = Failed induction/Failure to progress
  3. = Cord prolapse
  4. = Non-reassuring fetal tracing
  5. = Malpresentation
  6. = Placental abruption
  7. = Other
Time Frame: Induction to delivery
Population: Only 51 in the Combined arm and 53 in the single arm delivered by cesarean.
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Approach: Foley Balloon + Vaginal Misoprostol | Single Approach: Vaginal Misoprostol Only
Number analyzed (Participants) | 51 | 53
Participants
  Arrest disorders | 31 | 28
  Nonreassuring fetal heart rate | 13 | 18
  Other | 7 | 7

3. Secondary Outcome: Induction-to-delivery Interval in Hours
Time Frame: Induction to delivery
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Combined Approach: Foley Balloon + Vaginal Misoprostol | Single Approach: Vaginal Misoprostol Only
Number analyzed (Participants) | 113 | 123
hours | 24.8 (13.8) | 24.5 (14.0)

4. Secondary Outcome: Number of Participants With a Need for Oxytocin Augmentation
Time Frame: Induction to delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Approach: Foley Balloon + Vaginal Misoprostol | Single Approach: Vaginal Misoprostol Only
Number analyzed (Participants) | 113 | 123
Participants | 89 | 103

5. Secondary Outcome: Number of Participants Exhibiting Tachysystole Resulting in Fetal Heart Rate Abnormalities
Description: Uterine tachysystole is a condition of excessively frequent uterine contractions during pregnancy. Tachysystole is indicated ≥ 5 contractions in a 10 minute period averaged over a 30-minute window.
Time Frame: Induction to delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Approach: Foley Balloon + Vaginal Misoprostol | Single Approach: Vaginal Misoprostol Only
Number analyzed (Participants) | 113 | 123
Participants | 10 | 20

6. Secondary Outcome: Number of Participants With Clinical Chorioamnionitis
Description: Clinical chorioamnionitis is indicated by maternal fever ≥ 100.4 Fahrenheit, uterine fundal tenderness, maternal or fetal tachycardia (>100/min and >160/min, respectively), and purulent or foul amniotic fluid.
Time Frame: Induction to delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Approach: Foley Balloon + Vaginal Misoprostol | Single Approach: Vaginal Misoprostol Only
Number analyzed (Participants) | 113 | 123
Participants | 1 | 1

7. Secondary Outcome: Number of Participants With a Need for Operative Vaginal Delivery
Time Frame: Induction to delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Approach: Foley Balloon + Vaginal Misoprostol | Single Approach: Vaginal Misoprostol Only
Number analyzed (Participants) | 113 | 123
Participants | 5 | 6

8. Secondary Outcome: Composite Maternal Morbidity as Indicated by the Number of Participants With Measures of Maternal Morbidity
Description: Measures of maternal morbidity assessed:
  * Maternal ICU admission
  * Postpartum endometritis
  * Surgical-site infections prior to discharge
  * Venous thromboembolism
  * Need for transfusion
  * Maternal death
Time Frame: Induction to discharge (approximately 5 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Approach: Foley Balloon + Vaginal Misoprostol | Single Approach: Vaginal Misoprostol Only
Number analyzed (Participants) | 113 | 123
Participants
  Maternal ICU Admission | 0 | 3
  Postpartum endometritis | 3 | 0
  Surgical site infection | 5 | 1

9. Secondary Outcome: Number of Newborns Admitted to the Neonatal Intensive Care Unit (NICU)
Time Frame: From delivery to neonatal discharge (approximately 2 to 7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Approach: Foley Balloon + Vaginal Misoprostol | Single Approach: Vaginal Misoprostol Only
Number analyzed (Participants) | 113 | 123
Participants | 24 | 20

10. Secondary Outcome: Number of Newborns With Transient Tachypnea (TTN)
Time Frame: From delivery to neonatal discharge (approximately 2 to 7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Approach: Foley Balloon + Vaginal Misoprostol | Single Approach: Vaginal Misoprostol Only
Number analyzed (Participants) | 113 | 123
Participants | 5 | 5

11. Secondary Outcome: Number of Newborns With Respiratory Distress Syndrome (RDS)
Time Frame: From delivery to neonatal discharge (approximately 2 to 7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Approach: Foley Balloon + Vaginal Misoprostol | Single Approach: Vaginal Misoprostol Only
Number analyzed (Participants) | 113 | 123
Participants | 5 | 4

12. Secondary Outcome: Number of Newborns With Meconium Aspiration Syndrome
Time Frame: From delivery to neonatal discharge (approximately 2 to 7 days)
Population: Data was not collected for this outcome measure.
Arm/Group | Combined Approach: Foley Balloon + Vaginal Misoprostol | Single Approach: Vaginal Misoprostol Only
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Number of Newborns With Culture-proven Sepsis
Time Frame: From delivery to neonatal discharge (approximately 2 to 7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Approach: Foley Balloon + Vaginal Misoprostol | Single Approach: Vaginal Misoprostol Only
Number analyzed (Participants) | 113 | 123
Participants | 0 | 1

14. Secondary Outcome: Number of Newborns With Seizures
Time Frame: From delivery to neonatal discharge (approximately 2 to 7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Approach: Foley Balloon + Vaginal Misoprostol | Single Approach: Vaginal Misoprostol Only
Number analyzed (Participants) | 113 | 123
Participants | 0 | 0

15. Secondary Outcome: Composite Neonatal Morbidity as Indicated by the Number of Newborns With Measures of Neonatal Morbidity
Description: Measures of neonatal morbidity assessed:
  * Apgar score ≤ 7 at 5 mins
  * Umbilical cord potential of hydrogen (pH) < 7.1
  * Neonatal injury: brachial plexus injury, fracture
  * Perinatal death
Time Frame: From delivery to neonatal discharge (approximately 2 to 7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Approach: Foley Balloon + Vaginal Misoprostol | Single Approach: Vaginal Misoprostol Only
Number analyzed (Participants) | 113 | 123
Participants
  Apgar score < 7 at 5 minutes | 4 | 3
  cord pH < 7.1 | 5 | 5
  any neonatal injury | 3 | 3

ADVERSE EVENTS:
Time Frame: From time of induction to time of discharge (about 5 days for mothers, and about 3-8 days for infants)
Arm/Group | Combined Approach: Foley Balloon + Vaginal Misoprostol | Single Approach: Vaginal Misoprostol Only
All-Cause Mortality (participants affected / at risk) | 0/113 | 0/123
Serious Adverse Events (participants affected / at risk) | 0/113 | 0/123
Other Adverse Events (participants affected / at risk) | 0/113 | 0/123

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/29/NCT02639429/Prot_SAP_000.pdf